CLINICAL TRIAL: NCT03774485
Title: Longitudinal Study of Myoelectric GutPrint of Healthy Controls and Crohn's Disease Patients During Flare and Remission
Brief Title: Myoelectric GutPrint-Crohn's Disease
Acronym: Gutcheck-CD
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); G-Tech Corporation (Industry)
Responsible Party: Principal Investigator, Sidhartha Ranjit Sinha, Assistant Professor, Stanford University
Other Study IDs: IRB48539
Record Dates: First submitted 2018-11-29; First posted 2018-12-13 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls: Record gastrointestinal motility by G-Tech Gutcheck Myoelectric recording device in healthy controls. The investigator does not change the routine medical care of study participants.
  Interventions: Device: G-Tech Gutcheck Myoelectric recording device
- Crohn's disease (remission state): Record gastrointestinal motility by G-Tech Gutcheck Myoelectric recording device in subjects with Crohn's disease (remission state). The investigator does not change the routine medical care of study participants.
  Interventions: Device: G-Tech Gutcheck Myoelectric recording device
- Crohn's disease (flare state): Record gastrointestinal motility by G-Tech Gutcheck Myoelectric recording device in subjects with Crohn's disease (flare state). The investigator does not change the routine medical care of study participants.
  Interventions: Device: G-Tech Gutcheck Myoelectric recording device

INTERVENTIONS:
Device: G-Tech Gutcheck Myoelectric recording device — Three G-Tech patches are placed on the abdomen of the patient to record myoelectric activity.
  Other Names: Gastro-intestinal electrical recording

SUMMARY:
A feasibility study for assessing and recording myoelectric activity in patients for early detection of flare in patients with Crohn's disease and differentiating the myoelectric signals from Crohn's disease patients in remission state and healthy controls.

DETAILED DESCRIPTION:
Crohn's disease (CD) patients can have a chronic, relapsing course with frequent flares despite aggressive therapy. Flares are often difficult to predict. The goal of disease monitoring is to identify patients at risk for flare in order to treat earlier, with the hope of maintaining remission and avoiding irreversible bowel damage such as fistulas and strictures that may lead to surgery. Although endoscopic visualization of the mucosa allows in some cases ability to predict flare and determine deep remission, this procedure is invasive and requires anesthesia and a bowel preparation, and is not without risk. Abdominal pain, cramps and diarrhea are particularly common symptoms of CD, which are associated with alteration of gastrointestinal (GI) motility. Thus better understanding of GI motility patterns in CD flare and remission states may be helpful for prediction of flare for guiding appropriate therapy.

The goal of this study is to determine whether the motility patterns measured by the G-Tech non-invasive, wireless patch system can provide useful insight for routine CD care. Three G-Tech patches will be placed on the patients' abdomen and they will be given an iPod Touch to carry with them for the next 3-6 days. Data from the patches is processed offline to obtain motility patterns of the stomach, small intestine and colon. These patterns represent a rich trove of data that can be studied in multiple ways to provide comparisons and insight. Some examples are the overall strength of motor activity in each of the organs, the duration and rhythmicity, the correlation with meals, pain events and bowel movements, day to day variations and their correlation with symptoms, and diurnal effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease and healthy subjects above the age of 18 who are able to give consent and follow direction.

Exclusion Criteria:

* Patients or subjects under the age of 18, pregnant, and those unable to give consent or follow direction.
* Healthy subjects with gastrointestinal symptoms or history of gastrointestinal surgeries.
* Patients with severe Crohn's disease due to complexity of disease, complication, and potential needs for surgery.
* Patients with bowel surgeries due to potential impact on the G-Tech results. For similar reasons we will exclude patients on new medications (e.g. within 3 months of enrollment) known to alter GI motility but we will not exclude patients on stable doses or chronic GI motility agents as this mimics "real world" in which the G-Tech patch will be used and we can learn the stability of the motility recordings over time in stable patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects without gastrointestinal symptoms or history of gastrointestinal surgeries.
  Patients with Crohn's disease in remission state or flare state (exclude severe Crohn's disease due to complexity of disease, complication, and potential needs for surgery; on new medications 【e.g. within 3 months of enrollment】 known to alter GI motility or bowel surgeries due to potential impact on the G-Tech results)
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Myoelectric activity pattern (physiological parameters) | change from baseline at 1 month, 3 months and 6 months after recruitment
  Myoelectric activity pattern in Crohn's disease patients versus healthy controls

SECONDARY OUTCOMES:
Number of anticipated Adverse Events | Up to 6 days
  Device related anticipated adverse events; such as, skin irritation due to adhesive from the skin patch.
Number of unanticipated adverse device effects | Up to 6 days
  Unanticipated adverse device effects

CONTACTS AND LOCATIONS:
Overall Officials: Sidhartha Sinha, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
We will share the data through publication of results. Individual participant data was not promised to be shared.

REFERENCES:
- [Background] Dua MM, Navalgund A, Axelrod S, Axelrod L, Worth PJ, Norton JA, Poultsides GA, Triadafilopoulos G, Visser BC. Monitoring gastric myoelectric activity after pancreaticoduodenectomy for diet "readiness". Am J Physiol Gastrointest Liver Physiol. 2018 Nov 1;315(5):G743-G751. doi: 10.1152/ajpgi.00074.2018. Epub 2018 Jul 26. PMID 30048596
- [Background] Navalgund A, Axelrod S, Axelrod L, Singhal S, Tran K, Legha P, Triadafilopoulos G. Colon Myoelectric Activity Measured After Open Abdominal Surgery with a Noninvasive Wireless Patch System Predicts Time to First Flatus. J Gastrointest Surg. 2019 May;23(5):982-989. doi: 10.1007/s11605-018-4030-4. Epub 2018 Nov 2. PMID 30390183
- [Background] Xavier RJ, Podolsky DK. Unravelling the pathogenesis of inflammatory bowel disease. Nature. 2007 Jul 26;448(7152):427-34. doi: 10.1038/nature06005. PMID 17653185
- [Background] Schoepfer AM, Trummler M, Seeholzer P, Seibold-Schmid B, Seibold F. Discriminating IBD from IBS: comparison of the test performance of fecal markers, blood leukocytes, CRP, and IBD antibodies. Inflamm Bowel Dis. 2008 Jan;14(1):32-9. doi: 10.1002/ibd.20275. PMID 17924558
- [Background] Abdalla MI, Sandler RS, Kappelman MD, Martin CF, Chen W, Anton K, Long MD. Prevalence and Impact of Inflammatory Bowel Disease-Irritable Bowel Syndrome on Patient-reported Outcomes in CCFA Partners. Inflamm Bowel Dis. 2017 Feb;23(2):325-331. doi: 10.1097/MIB.0000000000001017. PMID 28092305
- [Background] Barratt SM, Leeds JS, Robinson K, Lobo AJ, McAlindon ME, Sanders DS. Prodromal irritable bowel syndrome may be responsible for delays in diagnosis in patients presenting with unrecognized Crohn's disease and celiac disease, but not ulcerative colitis. Dig Dis Sci. 2011 Nov;56(11):3270-5. doi: 10.1007/s10620-011-1783-y. Epub 2011 Jun 22. PMID 21695401
- [Background] Grover M, Herfarth H, Drossman DA. The functional-organic dichotomy: postinfectious irritable bowel syndrome and inflammatory bowel disease-irritable bowel syndrome. Clin Gastroenterol Hepatol. 2009 Jan;7(1):48-53. doi: 10.1016/j.cgh.2008.08.032. Epub 2008 Sep 3. PMID 18848909
- [Background] von Stein P, Lofberg R, Kuznetsov NV, Gielen AW, Persson JO, Sundberg R, Hellstrom K, Eriksson A, Befrits R, Ost A, von Stein OD. Multigene analysis can discriminate between ulcerative colitis, Crohn's disease, and irritable bowel syndrome. Gastroenterology. 2008 Jun;134(7):1869-81; quiz 2153-4. doi: 10.1053/j.gastro.2008.02.083. Epub 2008 Mar 2. PMID 18466904
- [Background] Minderhoud IM, Oldenburg B, Wismeijer JA, van Berge Henegouwen GP, Smout AJ. IBS-like symptoms in patients with inflammatory bowel disease in remission; relationships with quality of life and coping behavior. Dig Dis Sci. 2004 Mar;49(3):469-74. doi: 10.1023/b:ddas.0000020506.84248.f9. PMID 15139501
- [Background] Bickelhaupt S, Pazahr S, Chuck N, Blume I, Froehlich JM, Cattin R, Raible S, Bouquet H, Bill U, Rogler G, Frei P, Boss A, Patak MA. Crohn's disease: small bowel motility impairment correlates with inflammatory-related markers C-reactive protein and calprotectin. Neurogastroenterol Motil. 2013 Jun;25(6):467-73. doi: 10.1111/nmo.12088. Epub 2013 Mar 18. PMID 23495824
- [Background] Bickelhaupt S, Froehlich JM, Cattin R, Patuto N, Tutuian R, Wentz KU, Culmann JL, Raible S, Bouquet H, Bill U, Patak MA. Differentiation between active and chronic Crohn's disease using MRI small-bowel motility examinations - initial experience. Clin Radiol. 2013 Dec;68(12):1247-53. doi: 10.1016/j.crad.2013.06.024. Epub 2013 Aug 21. PMID 23973163